CLINICAL TRIAL: NCT03506711
Title: Non-invasive Assessment of Endothelial Function in Children and Adolescents With Type 1 Diabetes Mellitus Using Isometric Handgrip Exercise -MRI: A Feasibility Study
Brief Title: Isometric Handgrip Exercise -MRI in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Michael Hauschild, Head of clinical pediatric endocrinology diabetology unit, University of Lausanne Hospitals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CER-VD 213/15
Record Dates: First submitted 2018-03-16; First posted 2018-04-24 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Type 1 Diabetes Mellitus; Coronary Artery Disease
Keywords: Type 1 Diabetes Mellitus; MRI; Isometric handgrip exercise; Children; Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1DM Children and adolescents (Active Comparator): Children and adolescents with Type 1 Diabetes Mellitus
  Interventions: Diagnostic Test: Isometric Handgrip Exercise during magnetic resonance imaging
- Healthy Children and adolescents (Active Comparator): Healthy community-dwelling children on no medication
  Interventions: Diagnostic Test: Isometric Handgrip Exercise during magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Isometric Handgrip Exercise during magnetic resonance imaging — Coronary endothelial function are assessed by MRI with imaging studies done at baseline (at rest) and during IHE (under stress). Maximum grip strength is determined using an MRI-compatible dynamometer (Grip Force Fiber Optic Response Pad, Current Designs Inc., Philadelphia, USA) prior to baseline imaging.

SUMMARY:
This project aims to assess coronary vessel response to isometric handgrip exercise (IHE) during magnetic resonance imaging (MRI) in children with T1D children and healthy controls. The investigators will compare the groups in terms of surrogate markers of intima media alteration and arterial stiffness, i.e. carotid intima media thickness (CIMT) and aortic pulse wave velocity (PWV).

DETAILED DESCRIPTION:
Background Type 1 diabetes mellitus (T1D) in children and adolescents is associated with significant cardiovascular morbidity and mortality. Early detection of vascular dysfunction is key to management yet assessment is invasive - which is particularly challenging when considering pediatric patient populations. Recently, a novel approach using isometric handgrip exercise (IHE) during magnetic resonance imaging (MRI) has been developed to evaluate coronary endothelial function in adults.

This project aims to assess coronary vessel response to IHE using MRI in children with T1D children and healthy controls. In addition, the investigators will compare the groups in terms of surrogate markers of intima media alteration and arterial stiffness, i.e. carotid intima media thickness (CIMT) and aortic pulse wave velocity (PWV).

Community-dwelling healthy volunteers (<18 years-old) and children with type 1 diabetes mellitus (disease duration ≥ 5 years) are recruited. IHE-MRI studies are conducted and measurements are recorded at rest (baseline) and under stress (IHE at 30% maximal effort). Carotic Ultrasound and Sphygmocor CPV System are used to assess CIMT and PWV respectively. Student's T-tests are used to compare results between groups.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes mellitus or
* Healthy community-dwelling children on no medications

Exclusion Criteria:

* smoking
* obesity (BMI >97th percentile)
* systolic or diastolic hypertension (>90th percentile)
* inflammatory process.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in coronary cross sectional area (mm2) | Baseline and up to 3 years
  Change from rest to that during isometric handgrip exercise (IHE).

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Endocrinology, Diabetology and Obesity Unit, Service of Pediatrics, Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yerly J, Gubian D, Knebel JF, Schenk A, Chaptinel J, Ginami G, Stuber M. A phantom study to determine the theoretical accuracy and precision of radial MRI to measure cross-sectional area differences for the application of coronary endothelial function assessment. Magn Reson Med. 2018 Jan;79(1):108-120. doi: 10.1002/mrm.26646. Epub 2017 Mar 5. PMID 28261859
- [Background] Hays AG, Stuber M, Hirsch GA, Yu J, Schar M, Weiss RG, Gerstenblith G, Kelle S. Non-invasive detection of coronary endothelial response to sequential handgrip exercise in coronary artery disease patients and healthy adults. PLoS One. 2013;8(3):e58047. doi: 10.1371/journal.pone.0058047. Epub 2013 Mar 11. PMID 23536782